CLINICAL TRIAL: NCT01822184
Title: A Prospective, Longitudinal, Observational Study to Evaluate Neurodevelopmental Status in Pediatric Patients With Hunter Syndrome (MPS II)
Brief Title: Observational Study to Evaluate Neurodevelopmental Status in Pediatric Patients With Hunter Syndrome (MPS II)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-HIT-090
Record Dates: First submitted 2013-03-12; First posted 2013-04-02 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Mucopolysaccharidosis (MPS); Hunter Syndrome
Keywords: Neurodevelopmental Status; Pediatric Hunter syndrome patients; Central Nervous System (CNS) involvement; Observational study; Cognitive impairment
MeSH Terms: conditions — Mucopolysaccharidoses; Mucopolysaccharidosis II; Margins of Excision; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genotyping of the iduronate-2-sulfatase gene will be required ONLY for those patients who have not had a previous genotyping sample analysis performed at the selected diagnostic laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Observational non-treatment study

SUMMARY:
Hunter syndrome (Mucopolysaccharidosis II, [MPS II]) is a rare, genetically linked lysosomal storage disease (LSD) caused by deficiency of the enzyme, iduronate-2-sulfatase (I2S). Most MPS II patients will present with some degree of neurodevelopmental involvement, ranging from severe cognitive impairment and behavioral problems to mildly impaired cognition. This is an observational study; no investigational treatment will be administered. The primary objective of this study is to evaluate the neurodevelopmental status of pediatric patients with MPS II over time and to gain information to guide future treatment studies in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be considered eligible for enrollment:

1. a. The patient has a deficiency in iduronate-2-sulfatase enzyme activity AND b. The patient has a documented mutation in the iduronate-2-sulfatase gene. OR c. The patient has a normal enzyme activity level of one other sulfatase
2. The patient is male, and is at least 2 years of age and less than 18 years of age at the time of informed consent.
3. The patient must have sufficient auditory capacity at enrollment, with or without hearing aids, in the Investigator's judgment to complete the required protocol testing, and be compliant with wearing the aids on scheduled study visits.
4. The patient, patient's parent(s), or legally authorized guardian(s) has voluntarily signed an Institutional Review Board / Independent Ethics Committee-approved informed consent and/or assent form(s), as applicable.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. The patient has clinically significant non-Hunter syndrome-related CNS involvement or medical or psychiatric comorbidity(ies) which, in the investigator's judgment, may interfere with the accurate administration and interpretation of protocol assessments, affect study data, or confound the integrity of study results.
2. The patient has a general conceptual ability score (GCA) or a developmental quotient on the cognitive scale below 55 at Screening.
3. The patient is participating in an interventional clinical trial or has participated in an interventional clinical trial within 30 days prior to enrollment; participation in non interventional observational studies is permitted.

Ages: 2 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male MPS II patients between 2<18 years of age at time of informed consent
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental parameters of cognitive function over time in pediatric patients with MPS II | 24 months
Neurodevelopmental parameters of adaptive function over time in pediatric patients with MPS II | 24 months

SECONDARY OUTCOMES:
Reported adverse events | 24 months
  Type and severity measurements
Medication usage | 24 months
Quality of life | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- United States (3):
  - Childrens Hospital & Research Center Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of North Carolina Division of Genetics and Metabolism, Chapel Hill, North Carolina
- Hospital Universitario Austral, Pilar, Buenos Aires, Argentina
- Instituto Nacional De Pediatria, Mexico City, Mexico
- Hospital Infantil Universitario, Madrid, Spain
- Central Manchester University Hospitals NHS Foundation Trust Willink Biochemical Genetics Unit, St. Mary's Hospital, Manchester, M13 9WL, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Muenzer J, Burton BK, Amartino HM, Harmatz PR, Gutierrez-Solana LG, Ruiz-Garcia M, Wu Y, Merberg D, Alexanderian D, Jones SA. Neurodevelopmental status and adaptive behavior of pediatric patients with mucopolysaccharidosis II: a longitudinal observational study. Orphanet J Rare Dis. 2023 Nov 16;18(1):357. doi: 10.1186/s13023-023-02805-3. PMID 37974184
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fce4db2bf003ab4676a